CLINICAL TRIAL: NCT00983255
Title: A Double-Blind, Placebo-Controlled, Single & Multiple Ascending Dose, Safety, Tolerability, & PK Study of an IV Form of TR-701 Free Acid & an Open-Label, Crossover Absolute BA Determination of a TR-701 FA Tablet in Normal Healthy Adults
Brief Title: Ascending Dose Pharmacokinetic (PK) and Absolute Bioavailability (BA)
Acronym: IV/SAD/MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1986-008; TR701-107 (Other: TriusRX Unique ID)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Injections; tedizolid phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SAD/ Part A (Experimental): Single IV infusions of placebo or TR-701 FA given at 50, 100, 200, and 400 mg.
  Interventions: Drug: TR-701 FA for injection, 200 mg/vial
- MAD / Part B (Experimental): Multiple IV infusion of placebo or TR-701 FA given daily for 7 days at 200 and 400 mg.
  Interventions: Drug: TR-701 FA for injection, 200 mg/vial
- Bioavailability / Part C (Experimental): TR-701 FA tablet given once orally as a 200 mg tablet or TR-701 FA for injection given once as a 200 mg IV infusion.
  Interventions: Drug: TR-701 FA for injection, 200 mg/vial; Drug: TR-701 FA tablets
- Venous Tolerability/ Part D (Experimental): IV infusions of placebo and 200 mg TR-701 FA given daily for 3 days,
  Interventions: Drug: TR-701 FA for injection, 200 mg/vial

INTERVENTIONS:
Drug: TR-701 FA for injection, 200 mg/vial — TR-701 FA for injection will be given as a single infusion at doses of 50 mg, 100 mg, 200 mg, and 400 mg in SAD/Part A (Pilot and Cohorts 1 to 3). TR-701 FA for injection will be given as once daily infusions at doses of 200 mg and 400 mg for 7 days in MAD/Part B (Cohorts 4 & 5). TR-701 FA for injection will be given once as a 200 mg IV infusion in BA/Part C (Cohort 6). TR-701 FA 200 mg will be given daily for 3 days in Venous Tolerability/Part D
  Other Names: Torezolid Phospate
Drug: TR-701 FA tablets — TR-701 FA will be given once orally as a 200 mg tablet in Part C.
  Other Names: Torezolid Phosphate Tablet
  Arms: Bioavailability / Part C

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single rising and multiple rising IV doses of TR-701 FA and to determine the absolute bioavailability of oral TR-701 FA following single oral and IV dose administrations in healthy adult subjects.

DETAILED DESCRIPTION:
SAD/Part A.

* All subjects in the Pilot Cohort will receive a single infusion of 50 mg TR-701 FA for injection in 250 cc of saline over 180 minutes.
* Subjects in Cohort 1 will be randomized to receive a single infusion of placebo or 100 mg of TR-701 FA for injection in 250 or 500 cc of saline over 60 or 120 minutes.
* Subjects in Cohort 2 will be randomized to receive a single infusion of placebo or 200 mg of TR-701 FA for injection in 250 or 500 cc of saline over 60 or 120 minutes.
* Subjects in Cohort 3 will be randomized to receive a single infusion of placebo or 400 mg of TR-701 FA for injection in 250 or 500 cc of saline over 60 or 120 minutes.

MAD/Part B

* Subjects in Cohort 4 will be randomized to receive once daily infusions of placebo or 200 mg of TR-701 FA for injection in 250 cc of saline over 60 minutes for 7 days.
* Subjects in Cohort 5 will be randomized to receive once daily infusions of placebo or 300 mg of TR-701 FA for injection in 250 cc of saline over 60 minutes for 7 days.

BA/Part C

* Subjects in Cohort 6 will receive a single 60 minute infusion of 200 mg TR-701 FA for injection in 250 cc of saline and a singe oral dose of 200 mg TR-701 FA tablet in an open-label crossover design.

Venous Tolerability/Part D

- Subjects in Cohort 8 will receive once daily 60 minute infusions of 200 mg TR-701 FA for injection in 250 cc of saline for 3 days and once daily placebo infusions for 3 daysin a blinded crossover design.

ELIGIBILITY:
Inclusion Criteria:

* in good health
* body mass index of 20 to 29.9 kg/m2
* female subjects must be post menopausal for at least 1 year, surgically sterile, abstinent or agree to use an effective method of birth control

Exclusion Criteria:

* history or clinical manifestation of any clinically significant disorder
* history of hypersensitivity to any drug compound
* history of stomach or intestinal surgery or resection
* history of infections of unexplained frequency or severity
* history of alcoholism or drug addiction within 1 year
* use of any tobacco- or nicotine-containing products within 6 months
* use of alcohol-, grapefruit-, caffeine-, or high tyramine-containing foods or beverages
* use of any other medications
* pregnancy, lactation, or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety Assessments | 10 days

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of TR-701 and its microbiologically active moiety TR-700 after single and multiple IV doses of TR-701 FA | 10 days
To determine the absolute bioavailability of oral TR-701 FA following single oral and IV dose administrations in healthy adult subjects | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, MD, Principal Investigator — Covance Clinical Research Unit, Madison, WI, USA
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Flanagan S, Fang E, Munoz KA, Minassian SL, Prokocimer PG. Single- and multiple-dose pharmacokinetics and absolute bioavailability of tedizolid. Pharmacotherapy. 2014 Sep;34(9):891-900. doi: 10.1002/phar.1458. Epub 2014 Jul 3. PMID 24989138